CLINICAL TRIAL: NCT00986986
Title: Prospective Randomized Pilot Study of the Effect of Niaspan on Endothelial Function in HIV-infected Subjects With Low HDL Cholesterol Levels
Brief Title: Study of Niacin on Endothelial Function in HIV-infected Subjects With Low High Density Lipoprotein Cholesterol Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dominic Chow, Associate Professor of Medicine and Pediatrics, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDO; Department of Defense (Other Grant/Funding Number: 06187003)
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-07

CONDITIONS: HIV Infections; Dyslipidemia; Endothelial Dysfunction
Keywords: Human immunodeficiency virus; Low high density lipoprotein; Endothelial function; Flow-mediated vasodilation
MeSH Terms: conditions — HIV Infections; Dyslipidemias; Acquired Immunodeficiency Syndrome | interventions — Niacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Drug (extended release niacin) (Experimental): Subjects in this arm will be given 12 weeks of extended release niacin. Intervention: extended release niacin (Niaspan) starting at 500 mg by mouth daily and titrated to a maximum dose of 1500 mg by mouth daily. Titration will depend on patient tolerability.
  Interventions: Drug: extended release niacin
- Observation (No Intervention): Subjects in this arm will be monitored for 12 weeks and will not receive extended release niacin

INTERVENTIONS:
Drug: extended release niacin — Active arm subjects will start extended release niacin (Niaspan) at 500 mg per night (by mouth once a daily) and titrate to a maximum tolerated dose (not exceeding 1500 mg per night (by mouth once a day) for 12 weeks. Titration will depend on patient tolerability of Niaspan.
  Other Names: Niaspan
  Arms: Active Drug (extended release niacin)

SUMMARY:
This study is a pilot study examining the effect of extended-release niacin (Niaspan ®) on flow-mediated vasodilation (FMD) of the brachial artery, among human immunodeficiency virus (HIV)-1 infected individuals with low high density lipoprotein (HDL). Brachial artery diameter will be measured by high-resolution ultrasound at entry and week 12 of study. The primary comparisons will be change in FMD from baseline to 12 weeks within each of the two arms. The second specific aim will be to investigate the proportion of the effect of extended-release niacin on other known cardiovascular markers.

DETAILED DESCRIPTION:
Low high density lipoprotein (HDL) and a lipid pattern consistent with atherogenic dyslipidemia are also common in the human immunodeficiency virus (HIV)infected population and is likely due, in large part, to the chronic inflammatory effect of HIV infection per se. While highly active antiretroviral therapy (HAART) and the resultant reconstitution of the immune system might be expected to lead to improvement in this lipid profile, studies from our own research as well as others clearly demonstrate that such therapy fails to fully correct the low HDL pattern. This coronary artery disease (CAD) risk in the HIV population is then further compounded by the dyslipidemic effects of various protease inhibitors and other antiretroviral medications used to treat HIV.

Endothelial dysfunction is an early marker of atherosclerosis that can be determined non-invasively utilizing assessment of flow-mediated vasodilation (FMD) of the brachial artery, which may be analogous to blood flow through coronary arteries. Using this novel technology and HIV as a model of a chronic inflammatory state, we propose to determine if increasing HDL in subjects with low HDL but no LDL elevation may have potential beneficial effects. Our overall hypothesis for this pilot project is that increasing HDL levels in HIV-infected subjects with low HDL by the use of extended-release niacin over a 12 week period will lead to an identifiable improvement in endothelial function.

Specific Aim 1. To compare endothelial function, measured by flow-mediated vasodilation (FMD) of the brachial artery, among HIV-1 infected individuals with low high density lipoprotein (HDL) before and after treatment with extended-release niacin (Niaspan ®)

* Conduct a prospective randomized 12-week clinical trial on HIV-1 infected individuals with low HDL and normal low density lipoprotein levels who plan to continue their current anti-retroviral regimens
* Subjects will be randomized to either a treatment or control arm
* Subjects randomized to the treatment arm will receive extended-release niacin (Niaspan ®) starting at 500 mg per night and titrated to a maximum tolerated dose (not exceeding 1500 mg per night)
* Assess changes in FMD of the brachial artery using high-resolution ultrasound from baseline to week 12 (Total of 2 FMD assessments)
* Correlate changes in HDL with changes in FMD

Hypothesis to be tested:

Use of extended-release niacin will improve FMD among HIV-1 infected individuals with low HDL

* Following 12 weeks of therapy, subjects treated with extended-release niacin will show a 8% improvement in FMD compared to controls
* There will be a positive correlation between changes in HDL with changes in FMD

Specific Aim 2. To evaluate changes in lipid parameters, insulin sensitivity and cardiovascular risk markers with changes in FMD among the treatment and control arms

* Assess and compare changes in non-HDL lipid and lipoprotein parameters with changes in FMD among the two arms
* Assess and compare changes in insulin sensitivity by homeostasis model assessment (HOMA) with changes in FMD among the two arms
* Assess and compare changes in cardiovascular risk markers such as adhesion molecules and C-reactive protein with changes in FMD among the two arms

Hypothesis to be tested:

There will be a correlation between improvements in lipid, insulin sensitivity and cardiovascular risk markers and FMD in the extended niacin treatment arm

SIGNIFICANCE and RATIONALE: Low HDL cholesterol levels elevate CAD risk independent of low density lipoprotein (LDL) cholesterol levels. In association with high triglyceride levels and with small LDL particle size, low HDL is part of the syndrome of atherogenic dyslipidemia. This form of dyslipidemia is characteristic of the underlying dyslipidemia found in HIV-infected subjects, likely represents the consequences of chronic inflammatory changes due to HIV, and contributes substantively to the CAD risk in this population even without the added risk from dyslipidemic antiretroviral medications. Primary CAD preventive modalities may be warranted for patients in the HIV population as well as in the general population who manifest this type of dyslipidemia. Niacin is currently the best medication available to elevate HDL cholesterol levels. Thus, using the novel technique of assessing flow-mediated dilatation of the brachial artery, a pilot project is proposed to assess whether the use of extended release niacin will lead to short term improvement in endothelial function. If successful, this study may lay the foundation for further studies into the potential use of niacin for prevention of CAD in patients who are particularly at risk for CAD due to low HDL cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Documented HIV infection
* Subjects must have taken HAART 6 months prior to study entry and must be on stable HAART (no dose change to antiretroviral medications) for at least 30 days immediately prior to study entry
* HDL < 40 mg/dL • LDL < 130 mg/dL
* All subjects with reproductive potential should utilize adequate contraception for the duration of this study and for at least 12 weeks following permanent discontinuation of study treatment. Acceptable methods include male condom, female condom, diaphragm, or intra-uterine device (IUD)

Exclusion Criteria:

* Known cardiac disease
* Arrhythmia
* History of angina
* Uncontrolled hypertension
* Pregnancy
* Breast-feeding
* Medication known to influence vasodilatation such as nitrates, metformin, pioglitazone, and rosiglitazone
* Heavy use of vitamin supplements
* Diagnosis of diabetes mellitus
* Treatment with lipid-lowering drugs within 6 weeks prior to study
* Hemoglobin <9.0 mg/dL
* Absolute neutrophil count <750 cells/mm3
* Platelet count <75,000 platelets/ mm3
* Alanine aminotransferase (ALT or SGOT)/ aspartate aminotransferase (AST or SGPT) / alkaline phosphatase > 2.5 x upper limit of normal (ULN)
* Creatinine >1.5 x ULN
* Individuals with an infection or other medical illness requiring hospitalization within 14 days prior to study entry
* Individuals who have active alcohol or drug abuse which, in the investigator's opinion, is sufficient to prevent adequate compliance with study therapy and evaluations
* Prior history of hypersensitivity reaction to niacin or any other component of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominic C Chow, MD, Principal Investigator — University of Hawaii - Hawaii Center for AIDS
Locations (1):
- University of Hawaii - Hawaii Center for AIDS, Honolulu, Hawaii, United States

REFERENCES:
- [Result] Chow DC, Stein JH, Seto TB, Mitchell C, Sriratanaviriyakul N, Grandinetti A, Gerschenson M, Shiramizu B, Souza S, Shikuma C. Short-term effects of extended-release niacin on endothelial function in HIV-infected patients on stable antiretroviral therapy. AIDS. 2010 Apr 24;24(7):1019-23. doi: 10.1097/QAD.0b013e3283383016. PMID 20216298

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was through the University of Hawaii, Hawaii Center for AIDS
Groups:
- Active Drug (Extended Release Niacin): Subjects in this arm will be given 12 weeks of extended release niacin
Period: Overall Study
Arm/Group | Active Drug (Extended Release Niacin) | Observation
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Drug (Extended Release Niacin) | Observation | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.96 (11.60) | 47.72 (10.81) | 48.84 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow-mediated Vasodilation (FMD) From Baseline to Study Week 12
Description: Brachial arterial flow-mediated dilation (FMD), assessed by high-resolution ultrasonography, reflects endothelium-dependent vasodilator function. The primary outcome is the change in FMD from baseline to study week 12.
Time Frame: Two time points (baseline and study week 12)
Population: HIV infected patients with HDL-C < 40
Measure: Median (Inter-Quartile Range); unit: percentage change in FMD
Groups:
- Extended Release Niacin: HIV infected individuals receiving extended release niacin
Arm/Group | Extended Release Niacin | Observation
Number analyzed (Participants) | 10 | 9
percentage change in FMD | 6.36 [4.85 to 7.87] | 2.73 [0.95 to 4.51]

2. Secondary Outcome: High-density Lipoprotein Cholesterol (HDL) Change From Baseline to Study Week 12
Description: HDL, often referred to "Good cholesterol levels", will be obtained in both arms. HDL is a marker of coronary heart disease.
Time Frame: Two time points (baseline and study week 12)
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Active Drug (Extended Release Niacin) | Observation
Number analyzed (Participants) | 10 | 9
mg/dl | 42.0 [39.3 to 43.5] | 27.0 [24.0 to 39.0]

3. Primary Outcome: Flow Mediated Vasodilation
Description: Flow mediated vasodilation is a marker of endothelial function
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: percentage change in FMD
Arm/Group | Active Drug (Extended Release Niacin) | Observation
Number analyzed (Participants) | 10 | 9
percentage change in FMD | 4.51 [4.46 to 8.32] | 3.25 [1.95 to 4.85]

4. Secondary Outcome: HDL
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Active Drug (Extended Release Niacin) | Observation
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
* Small sample size
* Un-blinded pilot study
* Increase in HDL was less than predicted in a non-HIV infected population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes